CLINICAL TRIAL: NCT03105362
Title: Tolerability of an Amino Acid-based Oral Rehydration Solution in Children With Short Bowel Syndrome
Brief Title: Amino Acid-based Oral Rehydration Solution in Children With Short Bowel Syndrome
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Issues w/ sponsor and recruitment
Sponsor: Boston Children's Hospital (Other)
Collaborators: Entrinsic Bioscience Inc. (Industry)
Responsible Party: Principal Investigator, Christopher Duggan, Professor of Pediatrics, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-P00024854
Record Dates: First submitted 2017-03-24; First posted 2017-04-07 (Actual); Results first posted 2019-12-17 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Short Bowel Syndrome
Keywords: Oral Rehydration Solutions
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Open label single center pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amino Acid-ORS arm (Experimental): Patients consumed an amino acid based oral rehydration solution (enterade®) as part of their oral rehydration care plan. Enterade® oral rehydration solution volumes varied from patient to patient depending on baseline clinical need.
  Interventions: Dietary Supplement: Enterade® oral rehydration solution

INTERVENTIONS:
Dietary Supplement: Enterade® oral rehydration solution — Commercially available amino acid based oral rehydration solution

SUMMARY:
This study will assess the tolerability and palatability of an amino acid based oral rehydration solution (enterade®) compared to current oral rehydration solution among children with short bowel syndrome .

DETAILED DESCRIPTION:
Patients with short bowel syndrome (SBS) have a critical reduction of the gut mass/function that is below the minimum needed to absorb nutrients and fluids required for adequate homeostasis. There are limited data regarding the optimal choice for oral rehydration in the setting of SBS that can maximize fluid absorption in the setting of diarrhea with limited intestinal absorptive surface area. The investigators propose a preliminary open label single center study assessing tolerability and palatability of enterade® ( an amino acid (AA) based oral rehydrating solution (ORS)) and compare to baseline. Eligible patients with SBS will participate in a 14-day trial monitoring and measuring tolerability and palatability of an AA-ORS, enterade®, in addition to their regular diet.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with a diagnosis of short bowel syndrome (as defined by surgical therapy for congenital or acquired gastrointestinal disease) between the ages of 1-17
* Patients who are in intestinal continuity or with diverting ileostomy, jejunostomy
* Patients must be on a stable enteral nutrition regimen with oral rehydration fluids that are taken orally.
* Stable GI medication regimen (e.g., loperamide, cholestyramine, small bowel bacterial overgrowth (SBBO) regimen)

Exclusion Criteria:

* Patients receiving IV antibiotics within the previous 72h.
* Patients with a primary diagnosis of a motility disorder (e.g., chronic intestinal pseudo-obstruction) or epithelial cell disorder (e.g., microvillus inclusion disease)
* Malnourished (as defined by Weight/Height Z-score (WHZ) <-2)

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2018-01-20 (Actual); Study Completion 2018-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Duggan, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Freedman SB, Cho D, Boutis K, Stephens D, Schuh S. Assessing the palatability of oral rehydration solutions in school-aged children: a randomized crossover trial. Arch Pediatr Adolesc Med. 2010 Aug;164(8):696-702. doi: 10.1001/archpediatrics.2010.129. PMID 20679159
- [Background] Modi BP, Langer M, Ching YA, Valim C, Waterford SD, Iglesias J, Duro D, Lo C, Jaksic T, Duggan C. Improved survival in a multidisciplinary short bowel syndrome program. J Pediatr Surg. 2008 Jan;43(1):20-4. doi: 10.1016/j.jpedsurg.2007.09.014. PMID 18206449
- [Background] Gosselin KB, Duggan C. Enteral nutrition in the management of pediatric intestinal failure. J Pediatr. 2014 Dec;165(6):1085-90. doi: 10.1016/j.jpeds.2014.08.012. Epub 2014 Sep 18. No abstract available. PMID 25242686
- [Background] King CK, Glass R, Bresee JS, Duggan C; Centers for Disease Control and Prevention. Managing acute gastroenteritis among children: oral rehydration, maintenance, and nutritional therapy. MMWR Recomm Rep. 2003 Nov 21;52(RR-16):1-16. PMID 14627948
- [Background] Faruque AS, Mahalanabis D, Hamadani J, Hoque SS. Hypo-osmolar sucrose oral rehydration solutions in acute diarrhoea: a pilot study. Acta Paediatr. 1996 Oct;85(10):1247-8. doi: 10.1111/j.1651-2227.1996.tb18240.x. PMID 8922094
- [Background] World Health Organization. Oral rehydration salts (ORS): A new reduced osmolarity formulation. Geneva: WHO, 2002 Contract No.: September 23, 2002.
- [Background] Santosham M, Burns BA, Reid R, Letson GW, Duncan B, Powlesland JA, Foster S, Garrett S, Croll L, Nyunt Nyunt W, et al. Glycine-based oral rehydration solution: reassessment of safety and efficacy. J Pediatr. 1986 Nov;109(5):795-801. doi: 10.1016/s0022-3476(86)80696-5. PMID 3534198
- [Background] Lima AA, Carvalho GH, Figueiredo AA, Gifoni AR, Soares AM, Silva EA, Guerrant RL. Effects of an alanyl-glutamine-based oral rehydration and nutrition therapy solution on electrolyte and water absorption in a rat model of secretory diarrhea induced by cholera toxin. Nutrition. 2002 Jun;18(6):458-62. doi: 10.1016/s0899-9007(02)00775-x. PMID 12044816
- [Background] Nightingale JM. The Sir David Cuthbertson Medal Lecture. Clinical problems of a short bowel and their treatment. Proc Nutr Soc. 1994 Jul;53(2):373-91. doi: 10.1079/pns19940043. No abstract available. PMID 7972152
- [Background] Lennard-Jones JE. Oral rehydration solutions in short bowel syndrome. Clin Ther. 1990;12 Suppl A:129-37; discussion 138. PMID 2187606
- [Background] Nightingale J, Woodward JM; Small Bowel and Nutrition Committee of the British Society of Gastroenterology. Guidelines for management of patients with a short bowel. Gut. 2006 Aug;55 Suppl 4(Suppl 4):iv1-12. doi: 10.1136/gut.2006.091108. No abstract available. PMID 16837533
- [Background] Radlovic V, Lekovic Z, Radlovic N, Lukac M, Ristic D, Simic D, Bijelic M. Significance of the application of oral rehydration solution to maintain water and electrolyte balance in infants with ileostomy. Srp Arh Celok Lek. 2013 May-Jun;141(5-6):325-8. doi: 10.2298/sarh1306325r. PMID 23858801
- [Background] Yin L, Gupta R, Vaught L, Grosche A, Okunieff P, Vidyasagar S. An amino acid-based oral rehydration solution (AA-ORS) enhanced intestinal epithelial proliferation in mice exposed to radiation. Sci Rep. 2016 Nov 23;6:37220. doi: 10.1038/srep37220. PMID 27876791
- [Background] Ching YA, Modi BP, Jaksic T, Duggan C. High diagnostic yield of gastrointestinal endoscopy in children with intestinal failure. J Pediatr Surg. 2008 May;43(5):906-10. doi: 10.1016/j.jpedsurg.2007.12.037. PMID 18485964
- [Background] Duro D, Kalish LA, Johnston P, Jaksic T, McCarthy M, Martin C, Dunn JC, Brandt M, Nobuhara KK, Sylvester KG, Moss RL, Duggan C. Risk factors for intestinal failure in infants with necrotizing enterocolitis: a Glaser Pediatric Research Network study. J Pediatr. 2010 Aug;157(2):203-208.e1. doi: 10.1016/j.jpeds.2010.02.023. Epub 2010 May 6. PMID 20447649
- [Background] Hull MA, Jones BA, Zurakowski D, Raphael B, Lo C, Jaksic T, Duggan C. Low serum citrulline concentration correlates with catheter-related bloodstream infections in children with intestinal failure. JPEN J Parenter Enteral Nutr. 2011 Mar;35(2):181-7. doi: 10.1177/0148607110381406. PMID 21378247
- [Background] Squires RH, Duggan C, Teitelbaum DH, Wales PW, Balint J, Venick R, Rhee S, Sudan D, Mercer D, Martinez JA, Carter BA, Soden J, Horslen S, Rudolph JA, Kocoshis S, Superina R, Lawlor S, Haller T, Kurs-Lasky M, Belle SH; Pediatric Intestinal Failure Consortium. Natural history of pediatric intestinal failure: initial report from the Pediatric Intestinal Failure Consortium. J Pediatr. 2012 Oct;161(4):723-8.e2. doi: 10.1016/j.jpeds.2012.03.062. Epub 2012 May 11. PMID 22578586
- [Background] Khan FA, Squires RH, Litman HJ, Balint J, Carter BA, Fisher JG, Horslen SP, Jaksic T, Kocoshis S, Martinez JA, Mercer D, Rhee S, Rudolph JA, Soden J, Sudan D, Superina RA, Teitelbaum DH, Venick R, Wales PW, Duggan C; Pediatric Intestinal Failure Consortium. Predictors of Enteral Autonomy in Children with Intestinal Failure: A Multicenter Cohort Study. J Pediatr. 2015 Jul;167(1):29-34.e1. doi: 10.1016/j.jpeds.2015.03.040. Epub 2015 Apr 25. PMID 25917765
- [Background] Fullerton BS, Sparks EA, Hall AM, Duggan C, Jaksic T, Modi BP. Enteral autonomy, cirrhosis, and long term transplant-free survival in pediatric intestinal failure patients. J Pediatr Surg. 2016 Jan;51(1):96-100. doi: 10.1016/j.jpedsurg.2015.10.027. Epub 2015 Oct 23. PMID 26561248
- [Background] Fayad IM, Hashem M, Duggan C, Refat M, Bakir M, Fontaine O, Santosham M. Comparative efficacy of rice-based and glucose-based oral rehydration salts plus early reintroduction of food. Lancet. 1993 Sep 25;342(8874):772-5. doi: 10.1016/0140-6736(93)91540-3. PMID 8103876
- [Background] Santosham M, Fayad I, Abu Zikri M, Hussein A, Amponsah A, Duggan C, Hashem M, el Sady N, Abu Zikri M, Fontaine O. A double-blind clinical trial comparing World Health Organization oral rehydration solution with a reduced osmolarity solution containing equal amounts of sodium and glucose. J Pediatr. 1996 Jan;128(1):45-51. doi: 10.1016/s0022-3476(96)70426-2. PMID 8551420
- [Background] Duggan C, Lasche J, McCarty M, Mitchell K, Dershewitz R, Lerman SJ, Higham M, Radzevich A, Kleinman RE. Oral rehydration solution for acute diarrhea prevents subsequent unscheduled follow-up visits. Pediatrics. 1999 Sep;104(3):e29. doi: 10.1542/peds.104.3.e29. PMID 10469812
- [Background] Duggan C, Fontaine O, Pierce NF, Glass RI, Mahalanabis D, Alam NH, Bhan MK, Santosham M. Scientific rationale for a change in the composition of oral rehydration solution. JAMA. 2004 Jun 2;291(21):2628-31. doi: 10.1001/jama.291.21.2628. No abstract available. PMID 15173155
- Available data/document: Study Protocol — http://www.childrenshospital.org/research-and-innovation/research/research-administration/office-of-clinical-investigation — For further details contact Lissette Jimenez, MD Email: lissette.jimenez@childrens.harvard.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female patients with a diagnosis of short bowel syndrome (as defined by surgical therapy for congenital or acquired gastrointestinal disease), who were on a stable enteral nutrition regimen (oral rehydration fluids taken orally) between the ages of 1-17 were recruited from clinic.
Pre-assignment Details: No run-in or wash out period prior to participating in study.
Groups:
- AA ORS Arm: Patients consumed (orally) an amino acid (AA) based oral rehydration solution (ORS) (enterade®) for 2 weeks as part of their baseline enteral hydration needs.
Period: Overall Study
Arm/Group | AA ORS Arm
Started | 4
Completed 1 Week of Study | 4
Completed 2 Weeks of Study | 3
Completed 2 Week Questionaire | 2
Completed | 2
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- AA ORS Arm: Patients will consume commercially amino acid based oral rehydration solution (enterade®).
  Enterade® oral rehydration solution: Commercially available amino acid based oral rehydration solution
Arm/Group | AA ORS Arm
Number analyzed (Participants) | 4
Age, Continuous [Mean (Full Range); unit: years] | 2.6 [2 to 13]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4
Primary Short Bowel Syndrome Diagnosis [Count of Participants; unit: Participants] — Participant's primary medical diagnosis that led to diagnosis of Short Bowel Syndrome
  Participants
    Hirschsprungs Disease | 2
    In-utero Volvulus | 1
    Necrotizing enterocolitis | 1
Residual Small Bowel Length [Mean (Full Range); unit: centimeters (cm)] — Population: One study participant had an unknown bowel length
  centimeters (cm)
    number analyzed (Participants) | 3
    (all) | 83.3 [65 to 120]
Presence of ileostomy or jejunostomy [Count of Participants; unit: Participants] | 2

OUTCOME MEASURES:

1. Primary Outcome: Average Stool Output Difference (First Week v. Second Week) for Patients With Ostomy
Description: Ostomy output measured as milliliters per day. The mean of outputs where compared between week 1(day 1-7) and week 2 (day 8-14). The difference (of the means) between weeks were reported.
Time Frame: Total study duration14 days
Population: Participants consumed amino acid-based ORS (enterade)
Measure: Mean (Full Range); unit: mL/day
Groups:
- Primary Outcome: AA ORS arm-Stool Output in subjects w/ ostomy
Arm/Group | Primary Outcome
Number analyzed (Participants) | 1
mL/day | 50 [50 to 50]

2. Secondary Outcome: Tolerance: Reported Episodes of Abdominal Distension and Emesis
Description: Number of episodes reported of abdominal distension and emesis during study period
Time Frame: 14 days
Population: Participants consuming amino acid oral rehydration solution (enterade)
Measure: Number; unit: Episodes
Groups:
- Outcome Measure (2): AA ORS arm-Emesis and/or abdominal distension
Arm/Group | Outcome Measure (2)
Number analyzed (Participants) | 3
Episodes
  Reported episodes of Abdominal Distension | 0
  Reported episodes of Emesis | 0

3. Other Pre Specified Outcome: Palatability Rating of Amino Acid ORS (Enterade®) Compared to Baseline ORS
Description: Rating of enterade® taste was compared to previous "patient baseline" oral rehydration solution taste. We compared measurements using the facial hedonic method 100-mm visual analog scale (worst (0mm) and best taste(100mm)). We utilized the difference between two measurements: Day 0 (baseline ORS) and Day 14 (last study day of Amino Acid-ORS consumption). The difference was reported (Day 14 minus value at Day 0).
Time Frame: 14 days
Population: Participants consuming enterade (amino acid oral rehydration solution)
Measure: Mean (Full Range); unit: mm
Groups:
- Outcome Measure (3): AA ORS arm-Palatability Rating
Arm/Group | Outcome Measure (3)
Number analyzed (Participants) | 2
mm | 0 [0 to 0]

4. Primary Outcome: Average Stool Output Difference (First Week v. Second Week) for Patients in Intestinal Continuity
Description: Output was measured as frequency of stools per day. The mean output was compared between week 1(day 1-7) and week 2 (day 8-14). The difference (of the means) between weeks were reported.
Time Frame: Total study duration 14 days
Population: Participants consumed amino acid-based ORS (enterade)
Measure: Mean (Full Range); unit: Stools per day
Groups:
- Primary Outcome: AA ORS arm-Stool output for subjects in continuity
Arm/Group | Primary Outcome
Number analyzed (Participants) | 1
Stools per day | .3 [.3 to .3]

ADVERSE EVENTS:
Time Frame: Data monitoring for adverse events were collected for 2 weeks
Groups:
- AA ORS Arm: Participants consuming enterade (amino acid-oral rehydration solution)
Arm/Group | AA ORS Arm
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT03105362/Prot_SAP_000.pdf